CLINICAL TRIAL: NCT02200692
Title: Risk Factors for Allergic Transfusion Reactions in Patients Receiving Plasma Transfusion
Brief Title: Allergic Transfusion Reactions in Plasma Transfusion
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/607; REK 2014/607 (Other: REC West 2014/607)
Record Dates: First submitted 2014-06-27; First posted 2014-07-25 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Allergy; Transfusion Reaction
Keywords: plasma transfusion; allergic transfusion reaction; transfusion reaction; blood transfusion; Solvent detergent plasma
MeSH Terms: conditions — Hypersensitivity; Transfusion Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples from patients receiving plasma transfusion and samples from plasma units transfused.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- plasma transfusion: Patients receiving plasma transfusion.

SUMMARY:
Allergic transfusion reactions are a common complication of transfusion by blood components containing plasma. This study aims to investigate passive transfer of Immunoglobin E antibodies as a risk factor of allergic reactions to plasma transfusion by use of Solvent Detergent plasma.

DETAILED DESCRIPTION:
Prospective observation study, aiming to measure transfer of Immunoglobin E antibodies and other factors associated with allergic complications in patients receiving plasma transfusion. Samples from patients and plasma units will be investigated. Samples frozen until investigation. To assess biological relevance of findings, additional analysis of basophil reactivity will be performed and information on clinical allergy collected by use of a questionaire .

In-patients will be recruited if receiving plasma transfusion during surgery or if an allergic transfusion complication occurs.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving plasma transfusion

Exclusion Criteria:

- Patients not able to complete sampling procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving plasma transfusion, mainly in relation to cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2014-06; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in concentration of allergen specific Immunoglobin E antibodies | Baseline and up to 8 weeks
  Multiple measurements over time needed to describe clearance of antibodies. Baseline samples defined as sample drawn less than 7 days before transfusion. After transfusion samples will be investigated daily during hospital stay (anticipated up to 14 days), and 4, 6 and/or 8 weeks after transfusion.

SECONDARY OUTCOMES:
Change from baseline in basophil reactivity measured by flow cytometry | Baseline and up to 8 weeks
  Multiple measurements over time needed to describe clearance of antibodies. Baseline samples defined as sample drawn less than 7 days before transfusion. After transfusion samples will be investigated during hospital stay, and 4, 6 and/or 8 weeks after transfusion.

OTHER OUTCOMES:
Number of patients with Serious and Non-Serious Adverse Events | Up to 8 weeks after transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Torunn O Apelseth, MD, PhD, Principal Investigator — Helse Bergen HF, Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No